CLINICAL TRIAL: NCT01520805
Title: A Phase 2a Open-Label Clinical Trial Evaluating Efficacy & Safety of CPI-613 in Patients With Refractory/Relapsed Acute Myeloid Leukemia (AML), and in Patients With Myelodysplastic Syndrome (MDS) Who Failed Hypomethylating Agents
Brief Title: Safety and Effectiveness Study of CPI-613 to Treat Refractory or Relapsed Leukemia and Myelodysplastic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-CPI-613-022; CL-CPI-613-022 (Other: Protocol Number)
Record Dates: First submitted 2012-01-20; First posted 2012-01-30 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: acute myeloid leukemia; myelodysplastic syndrome; refractory; relapsed; hypomethylating agents
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPI-613 (Experimental): CPI-613 will be intravenously infused over 2 hours, given twice weekly for 3 weeks followed by a week of rest.
  Interventions: Drug: CPI-613

INTERVENTIONS:
Drug: CPI-613 — CPI-613 drug product, provided in concentrated form at 50 mg/mL, must be diluted with D5W prior to administration. CPI-613 is to be infused intravenously (IV) via a central venous catheter. The dose of CPI-613 will be either the Maximum Tolerated Dose (MTD) or the highest No-Significant- Adverse-Effects-Dose-Level (NOAEL), as determined from the nearly completed Phase 1 dose-escalation clinical trial in patients with hematologic malignancies (i.e., Cornerstone Study# CL-CPI-613-009 or Wake Forest Study# CCCWFU 29109, under IND 107,800).
  Other Names: 6,8-bis-benzylsulfanyloctanoic acid; 6,8-bis(benzylthio)octanoic acid; 6,8-bis-benzylsulfonyloctanoic acid; Bylantra

SUMMARY:
The purpose of this study is to determine whether CPI-613 is effective and safe in either patients with refractory or relapsed acute myeloid leukemia (AML) or patients with myelodysplastic syndrome (MDS) who have failed therapy with a hypomethylating agent (such as decitabine [Vidaza] and azacitidine [AZA]).

DETAILED DESCRIPTION:
A new therapy for AML is necessary because, although there are several treatment options for patients with AML, these treatments are very toxic and not available to all AML patients or only useful for acute promyelocytic leukemia (APL). Also, there is essentially no treatment for patients with refractory or relapsed AML outside of bone marrow transplant. Accordingly, there is a great medical need for a safe and effective therapy for AML, especially refractory and relapsed AML. Also, although hypomethylating agents have been found to be effective against MDS, these agents are toxic. Furthermore, after relapsing from a hypomethylating agent, there is no treatment for this disease.

A nearly completed clinical trial of CPI-613 (Cornerstone Study# CL-CPI-613-009 or Wake Forest Study# CCCWFU 29109, under IND# 107,800) shows that CPI-613 is well tolerated at doses as high as 3,000 mg/m2. Results from this nearly completed trial also suggest that CPI- 613 may be effective against refractory and relapsed AML, as well as against MDS that is relapsed from a hypomethylating agent. Therefore, CPI-613 may be a suitable treatment option for refractory/relapsed AML and MDS relapsed from a hypomethylating agent. The promising preliminary efficacy data from Study# CL-CPI-613-009 (Wake Forest Study# CCCWFU 29109, under IND# 107,800) is the basis on which Cornerstone is conducting the current Phase 2a trial to further assess the efficacy of CPI-613 against these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Have either documented refractory or relapsed AML, or documented MDS of any risk group that has failed a hypomethylating agent (such as decitabine [Vidaza] and azacitidine [AZA]). (Therapy failure with a hypomethylating agent is defined as patients who have been sufficiently treated with hypomethylating agents without response in the opinion of the treating physician, or whose disease has progressed or relapsed while on a hypomethylating agent.) Has never been treated with CPI-613.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Expected survival >2 months.
* 18 years of age and older of both genders.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive, or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
* No radiotherapy, surgery or hormonal therapy for any kind of within 2 weeks prior to participating in this study. Patients must have fully recovered from the acute toxicities of any prior treatment with any anti-cancer drugs (including hypomethylating agents in MDS patients), radiotherapy or other anti-cancer modalities (i.e., returned to baseline status as noted before most recent treatment) for any tumors. Patients with persisting, stable chronic toxicities from such prior treatment ≤Grade 1 are eligible, but must be documented as such.
* Recombinant erythropoietin or G-CSF is not allowed, since CPI-613 does not induce myelosuppression.
* No evidence of active or serious infection of any kind within the past month. No systemic fungal, bacterial, viral or other infection not controlled, defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment.
* Signed informed consent form.

Exclusion Criteria:

* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity.
* Active heart disease including myocardial infarction within the previous 6 months, symptomatic coronary artery disease, abnormal ECG, or symptomatic congestive heart failure.
* Any active uncontrolled bleeding, or any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
* Dyspnea with minimal to moderate exertion. Patients with large pleural, pericardial, or peritoneal effusions.
* Evidence of active infection, or serious infection within the past month.
* Patients with active central nervous system (CNS) or epidural solid or hematologic tumors.
* Patients receiving any standard or investigational therapy for any tumor indication within the past 2 weeks, or any investigational agent for any indication within the past 4 weeks, prior to the study.
* Patients who have received immunotherapy of any type for any indications within the past 4 weeks prior to the study.
* Ongoing oral corticosteroids are not permitted. However, topical and inhaled corticosteroids are permitted, and prophylactic steroids are allowed for transfusion reactions.
* Life expectancy less than 2 months.
* Pregnant women, or women of child-bearing potential not using reliable means of contraception.
* Lactating females.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Unwillingness or inability to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Monitored until participants passed away, for an expected average of 6 months.

SECONDARY OUTCOMES:
Overall Remission Rate | Monitored at the end of every 4-week treatment cycle during treatment with CPI-613, for an expected average of 20 weeks.
Response Rate | Monitored at the end of every 4-week treatment cycle during treatment with CPI-613, for an expected average of 20 weeks.
Duration of Overall Remission | Monitored at the end of every 4-week treatment cycle during treatment with CPI-613, for an expected average of 20 weeks.
Progression Free Survival (PFS) | Monitored during treatment with CPI-613 and until participants passed away, which will be an expected average of 6 months.
Quality of Life (QOL) | Monitored before, during and 1 week after treatment with CPI-613, for an expected average of 20 weeks.
Safety | Monitored at the end of every 4-week treatment cycle during treatment with CPI-613, for an expected average of 20 weeks.
  Safety assessment will be based on clinical signs, vital signs, blood work, adverse events, AEs, etc.

CONTACTS AND LOCATIONS:
Overall Officials: King C Lee, Ph.D., Study Director — Cornerstone Pharmaceuticals
Locations (1):
- Cornerstone Pharmaceuticals, Inc, Cranbury, New Jersey, United States